CLINICAL TRIAL: NCT07103499
Title: Effects of Abdominal Endurance and Core Stabilization Exercises on Respiratory Functions in Overweight and Obese Women
Brief Title: Abdominal and Core Exercises on Respiratory Functions in Obese and Overweight Women (COREBREATH)
Acronym: COREBREATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, Ass.Prof., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/345
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Overweight; Pulmonary Disease; Muscle Weakness
Keywords: Obesity; Overweight; Pulmonary Function; Pilates; Core Stabilization; Abdominal Endurance; Breathing Exercises; Body Mass Index; Respiratory Rate
MeSH Terms: conditions — Obesity; Overweight; Lung Diseases; Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will participate in an 8-week supervised Pilates-based exercise program focused on core stabilization and abdominal endurance. Sessions will be held three times a week at Easyfiz Clinic using reformer and cadillac Pilates equipment. Each session will include diaphragmatic breathing-based warm-up and cool-down components.
  Interventions: Behavioral: Pilates-Based Core and Breathing Exercise Program
- Control Group (No Intervention): Participants in this group will not receive any specific exercise or breathing intervention. They will be instructed to maintain their usual daily activities during the study period.

INTERVENTIONS:
Behavioral: Pilates-Based Core and Breathing Exercise Program — An 8-week supervised Pilates-based exercise program for overweight and obese women, focusing on abdominal endurance and core stabilization. Sessions (3/week) include diaphragmatic breathing, use of reformer and cadillac equipment, and structured warm-up, main, and cool-down phases.
  Arms: Intervention Group

SUMMARY:
This study aims to examine the effects of an 8-week Pilates-based exercise program on breathing functions in overweight and obese women (BMI ≥ 25). The program includes exercises for abdominal endurance and core stabilization, performed three times a week.

Participants will be divided into two groups: an exercise group and a control group. Before and after the program, measurements will include lung function (spirometry), breathing rate, breath-holding time, abdominal mobility, core endurance (curl-up test), and quality of life (SF-36 questionnaire).

The goal is to find out whether this type of exercise can improve breathing and overall health in women with excess weight.

DETAILED DESCRIPTION:
This study aims to investigate the effect of an 8-week Pilates-based abdominal endurance and core stabilization exercise program on respiratory function in obese and overweight women (BMI ≥ 25). The intervention program is planned to last for a total of 24 sessions, 3 days a week. The exercises will be performed using reformer and cadillac devices, under the supervision of a physical therapist, at the Easyfiz Healthy Living Center.

Participants will be randomly assigned to two groups: an experimental group receiving the exercise intervention and a control group not receiving the intervention. Assessments conducted before and after the study for both groups will include the following parameters:

* Spirometry (FEV₁, FVC, FEV₁/FVC ratio),
* Respiratory rate,
* Breath-holding time (in seconds),
* Thoracoabdominal expansion (measured with a tape measure at the epigastric, subcostal, and lower costal levels),
* Core muscle endurance (using the ACSM Curl-Up test),
* Quality of life (using the 36-item Short Form - SF-36).

The exercise program will be planned in three phases:

Weeks 1-2: beginner level, Weeks 3-5: intermediate level, Weeks 6-8: advanced level. Each session will last approximately 45-50 minutes and will consist of a warm-up (diaphragmatic breathing and mobilization), main exercise (core stability and breathing-focused movements), and cool-down (stretching and breathing relaxation exercises).

This study aims to contribute to the field of cardiopulmonary rehabilitation by demonstrating the effects of a comprehensive exercise approach aimed at improving respiratory function and quality of life in obese individuals.

ELIGIBILITY:
inclusion criteria

1. Women aged 18-60
2. Body mass index (BMI) ≥ 25 kg/m² (obese and overweight)
3. Baseline FEV0 value ≥ 80% (measured by spirometry)
4. Individuals without respiratory disease (no diagnosis of asthma, COPD, etc.)
5. Individuals who have not engaged in regular exercise in the past 6 months
6. Individuals without orthopedic or neurological conditions that physically prevent participation in the exercise protocol
7. Non-pregnant individuals
8. Individuals who voluntarily agree to participate in the study and sign the informed consent form exclusion criteria

1. Individuals with a FEV0 value <80% (due to risk of obstructive lung disease) 2. Individuals who have undergone surgery in the abdomen, waist, or pelvic area within the last 6 months 3. Individuals with orthopedic, neurological, or systemic diseases that would prevent them from exercising 4. Individuals who have been engaging in regular exercise for 3 or more days per week in the past 3 months 5. Individuals with diagnosed respiratory diseases (e.g., asthma, COPD, etc.) 6. Individuals who are unable to comply with the exercise program due to psychiatric diagnosis or communication difficulties

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — woman
Enrollment: 48 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) - Spirometry | Baseline and at 8 weeks after the intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayıs Üniversitesi, Samsun, Atakum
  - Fizyoterapist Reyhan Arzum Apraş Özel Sağlık Meslek Hizmet Birimi, Çorum, Merkez

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.

REFERENCES:
- [Background] Souza C, Kruger RL, Schmit EFD, Wagner Neto ES, Reischak-Oliveira A, de Sa CKC, Loss JF. Cardiorespiratory Adaptation to Pilates Training. Res Q Exerc Sport. 2021 Sep;92(3):453-459. doi: 10.1080/02701367.2020.1749222. Epub 2020 Jun 4. PMID 32493165
- [Background] Afsari, Z., Rahimi, N. M., & Azimkhani, A. (2024). Investigating the Effects of Dynamic Neuromuscular Stabilization Exercises on Chest Mobility, Upright Sitting Height, and Quality of Life in Obese Women. Physical Treatments-Specific Physical Therapy Journal, 14(2), 137-146.